CLINICAL TRIAL: NCT05132504
Title: Phase II Study of Neoadjuvant Folfirinox Chemotherapy Followed by Pembrolizumab Followed by Surgery for Patients With Localized, Resectable Adenocarcinoma of the Pancreas
Brief Title: Neoadjuvant Folfirinox Combined With Pembrolizumab Followed by Surgery for Patients With Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ernest Ramsay Camp, Professor and Chief, Division of Surgical Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-50168
Record Dates: First submitted 2021-10-27; First posted 2021-11-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pembrolizumab; pancreatic cancer; pancreas adenocarcinoma; folfirinox
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Folfirinox and Pembrolizumab followed by sx for patients with pancreatic cancer (Experimental): Patients will receive 6 cycles of Folfirinox (Oxaliplatin 85 mg/m2, Leucovorin 400 mg/m2, Irinotecan 150 mg/m2, 5-Fluorouracil 2,400 mg/m2) with 2 cycles of Pembrolizumab 400 mg before surgical resection. Following surgery patients will receive 5-Fluorouracil based chemotherapy for up to 6 cycles with 7 more cycles of Pembrolizumab. Patients will receive a total of 9 doses of Q6week cycles of Pembrolizumab.
  Interventions: Drug: Pembrolizumab; Drug: Folfirinox

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be initiated starting with the Cycle 2 Day 1 and will be administered every 6 weeks with a max amount of 9 cycles throughout the study.
  Other Names: keytruda
Drug: Folfirinox — Once eligibility has been confirmed and the patient has been registered to the study, the patient will begin induction modified FOLFIRINOX (Oxaliplatin, Leucovorin, Irinotecan, 5-Fluorouracil) chemotherapy treatment. Each cycle is 14 days; a total of six cycles will be administered. Patients will receive growth factor support at the discretion of treating physician.
  Other Names: mFolfirinox

SUMMARY:
Abbreviated Title: Neoadjuvant FOLFIRINOX combined with Pembrolizumab followed by surgery for patients with resectable pancreatic cancer Trial Phase: Phase II Clinical Indication: Pancreatic ductal adenocarcinoma; Adenocarcinoma; AJCC I, II, or III; 1st Line neoadjuvant Trial Type: Interventional prospective Type of control: Historical Route of administration: IV Treatment Groups: Neoadjuvant FOLFIRINOX combined with Pembrolizumab followed by surgery for patients with resectable pancreatic cancer Number of trial participants: 30 Estimated enrollment period: 24 months Estimated duration of trial: 3.5 Years Duration of Participation:16 months Estimated average length of treatment per patient: 16 months

DETAILED DESCRIPTION:
This is a Phase II trial of NEOADJUVANT FOLFIRINOX CHEMOTHERAPY WITH PEMBROLIZUMAB followed by SURGERY and Adjuvant PEMBROLIZUMAB for Patients with LOCALIZED, RESECTABLE Adenocarcinoma of the pancreas. Investigators hypothesize that appropriately timed neoadjuvant FOLFIRINOX with anti-PD-1 mAb (pembrolizumab) can be administered safely and feasibly, and that this combination will lead to improved clinical response associated with enhanced numbers of immune cells in surgically resected pancreatic tumors. Patients will receive 6 cycles of FOLFIRINOX with 2 cycles of PEMBROLIZUMAB before surgical resection. Following surgery patients will receive 5FU based chemotherapy for up to 6 cycles with 7 more cycles of PEMBROLIZUMAB. Patients will receive a total of 9 doses of Q6week cycles of PEMBROLIZUMAB.

Toxicities will be continuously monitored using the method proposed by Ivanova et al. [Ivanova, A., Qaqish, B.F., and Schell, M.J. (2005). Continuous toxicity monitoring in phase II trials in oncology. Biometrics 61: 540-545.]. The method generates a Pocock-type stopping boundary for repeated testing for toxicity. Sequential boundaries will be used to monitor dose-limiting toxicity rate. The accrual will be halted if excessive numbers of dose-limiting toxicities are seen, that is, if the number of dose-limiting toxicities is equal to or exceeds boundary number out of the number of patients with full follow-up. This is a Pocock-type stopping boundary that yields the probability of crossing the boundary at most 5% when the rate of dose-limiting toxicity is equal to the acceptable rate of 25%.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age and has histologically or cytologically confirmed localized adenocarcinoma of the pancreas that is potentially resectable. Patients with islet cell or other neuroendocrine neoplasms are excluded.
2. Definition of localized, potentially resectable disease: a) Adequate CT or MRI to determine staging and eligibility based on radiologic interpretation. b) No extension to superior mesenteric artery (SMA) and hepatic artery. Patent superior mesenteric vein/portal vein (SMV/PV) with < 180-degree abutment and no evidence of invasion. c) Clear fat plane between the SMA and celiac axis. d) No extension to celiac axis and hepatic artery. e) Patent superior mesenteric vein and portal vein. f) No evidence of distant metastatic disease 3. If a female patient is of childbearing potential, she must have a negative urine pregnancy test documented within 72 hours of first intervention. 4. Fertile participants must use contraception considered adequate and appropriate as stated in Appendix 3 (pages 61-62).

5. Male participants: A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 220 days after the last dose of study treatment and refrain from donating sperm during this period.

6. Patient must not have received prior chemotherapy or radiation for pancreatic cancer. 7. Patient has an ECOG performance status PS 0-1. 8. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form before participation in any study-related activities.

9. A female participant is eligible to participate if:

a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 (pages 61-62). OR b. A WOCBP who is not pregnant, not breastfeeding, and agreeing to use proper contraception defined by the protocol (Appendix 3 [pages 61 - 62] and Table 18 [page 63]) for at least 160 days after the last dose of study treatment.

10. Have adequate organ function as defined in the following table (Table 3). Specimens must be collected within 14 days before the start of interventions.

Hematological Absolute neutrophil count (ANC) ≥1500/μL Platelets ≥100 000/μL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Renal Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Patient has borderline resectable, locally advanced unresectable, or advanced metastatic disease. Patients with neuroendocrine tumors, adenosquamous cancer, lymphoma of the pancreas, or ampullary cancer are also ineligible.
2. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
3. Patient has known infection with HIV.
4. Patient has undergone major surgery, other than diagnostic surgery (-e.g. diagnostic laparoscopy or placement of a central venous catheter), within 4 weeks before registration.
5. Patient has a history of allergy or hypersensitivity to the study drugs.
6. Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive chemotherapy and/or radiation therapy.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Patient has had clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before registration.
9. Patient is unwilling or unable to comply with study procedures.
10. Patient is enrolled in any other therapeutic clinical protocol or investigational trial.
11. Patients aged ≥ 80 are not excluded. However, candidates in this age group should be thoroughly evaluated before registration in the study, to ensure they are fit to receive chemotherapy, and to potentially undergo pancreaticoduodenectomy. In addition to meeting all of the baseline patient selection criteria, clinical judgment on their susceptibility to infection and expected stability of their performance status and suitability to receive intensive chemotherapy cycles, should be paid special attention to. Patients should not be enrolled in the study should there be any hesitation on any of these considerations. Baseline criteria for all patients enrolled in the study must be carefully evaluated and all criteria followed appropriately.
12. Patient has evidence of peripheral neuropathy Grade 2 or higher.
13. A WOCBP who has a positive urine pregnancy test within 72 hours prior to first intervention (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a second urine pregnancy test will be required. In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another urine pregnancy test must be performed and must be negative in order for the subject to start receiving study medication.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
15. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug.
16. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
17. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
18. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
19. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
20. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detectable HCV by RNA) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authorities.
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Determine if the neoadjuvant FOLFIRINOX chemotherapy followed by pembrolizumab followed by surgery will improve the overall response rate (ORR) for patients with localized, resectable adenocarcinoma of the pancreas. | 3 years
  The primary endpoints are overall response rate (ORR) defined as the proportion of patients with pathologic CR or PR. The primary analysis will compare the observed ORR to the null proportion of 5% using an exact binomial test.
  In addition, the percentage of ORR for the intervention with its 95% confidence interval will be presented.

SECONDARY OUTCOMES:
Estimate the effect of combination neoadjuvant therapy on the R0 resection rate | 3 years
  The percentage of R0 resection will be estimated with its 95% confidence interval.
Determine if the addition of pembrolizumab to neoadjuvant mFOLFIRINOX leads to improved CD8+ T cell frequencies in resected tumor samples in comparison to archived matched controls from patients meeting the same I/E criteria as those in the study. | 3 years
  Descriptive statistics will be provided. Group comparisons of CD8+ T cell frequencies will be performed.
Estimate the effect of combined neoadjuvant therapy on relapse-free survival, time to recurrence and overall survival. | 3 years
  Survival outcomes will be summarized with related 95% confidence interval.
Report of safety profile | 3 years
  This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for toxicity and Serious Adverse Event reporting, with the exception of skin- or nail-related toxicities, which will be graded using CTCAE version 5.0 with modifications.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest R. Camp, M.D., M.S.C.R., F.A.C.S., Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center (BSLMC)., Houston, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Macedo FI, Ryon E, Maithel SK, Lee RM, Kooby DA, Fields RC, Hawkins WG, Williams G, Maduekwe U, Kim HJ, Ahmad SA, Patel SH, Abbott DE, Schwartz P, Weber SM, Scoggins CR, Martin RCG, Dudeja V, Franceschi D, Livingstone AS, Merchant NB. Survival Outcomes Associated With Clinical and Pathological Response Following Neoadjuvant FOLFIRINOX or Gemcitabine/Nab-Paclitaxel Chemotherapy in Resected Pancreatic Cancer. Ann Surg. 2019 Sep;270(3):400-413. doi: 10.1097/SLA.0000000000003468. PMID 31283563
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Katz MH, Pisters PW, Lee JE, Fleming JB. Borderline resectable pancreatic cancer: what have we learned and where do we go from here? Ann Surg Oncol. 2011 Mar;18(3):608-10. doi: 10.1245/s10434-010-1460-y. No abstract available. PMID 21136179
- [Background] VanHouten JP, White RR, Jackson GP. A decision model of therapy for potentially resectable pancreatic cancer. J Surg Res. 2012 May 15;174(2):222-30. doi: 10.1016/j.jss.2011.08.022. Epub 2011 Sep 12. PMID 22079845
- [Background] Ghaneh P, Smith R, Tudor-Smith C, Raraty M, Neoptolemos JP. Neoadjuvant and adjuvant strategies for pancreatic cancer. Eur J Surg Oncol. 2008 Mar;34(3):297-305. doi: 10.1016/j.ejso.2007.07.204. Epub 2007 Oct 22. PMID 17936564
- [Background] Kircher SM, Krantz SB, Nimeiri HS, Mulcahy MF, Munshi HG, Benson AB 3rd. Therapy of locally advanced pancreatic adenocarcinoma: unresectable and borderline patients. Expert Rev Anticancer Ther. 2011 Oct;11(10):1555-65. doi: 10.1586/era.11.125. PMID 21999129
- [Background] Gillen S, Schuster T, Meyer Zum Buschenfelde C, Friess H, Kleeff J. Preoperative/neoadjuvant therapy in pancreatic cancer: a systematic review and meta-analysis of response and resection percentages. PLoS Med. 2010 Apr 20;7(4):e1000267. doi: 10.1371/journal.pmed.1000267. PMID 20422030
- [Background] Evans DB, Varadhachary GR, Crane CH, Sun CC, Lee JE, Pisters PW, Vauthey JN, Wang H, Cleary KR, Staerkel GA, Charnsangavej C, Lano EA, Ho L, Lenzi R, Abbruzzese JL, Wolff RA. Preoperative gemcitabine-based chemoradiation for patients with resectable adenocarcinoma of the pancreatic head. J Clin Oncol. 2008 Jul 20;26(21):3496-502. doi: 10.1200/JCO.2007.15.8634. PMID 18640930
- [Background] Kieler M, Unseld M, Bianconi D, Prager G. Challenges and Perspectives for Immunotherapy in Adenocarcinoma of the Pancreas: The Cancer Immunity Cycle. Pancreas. 2018 Feb;47(2):142-157. doi: 10.1097/MPA.0000000000000970. PMID 29346215
- [Background] Dosset M, Vargas TR, Lagrange A, Boidot R, Vegran F, Roussey A, Chalmin F, Dondaine L, Paul C, Lauret Marie-Joseph E, Martin F, Ryffel B, Borg C, Adotevi O, Ghiringhelli F, Apetoh L. PD-1/PD-L1 pathway: an adaptive immune resistance mechanism to immunogenic chemotherapy in colorectal cancer. Oncoimmunology. 2018 Mar 15;7(6):e1433981. doi: 10.1080/2162402X.2018.1433981. eCollection 2018. PMID 29872568
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Hackert T, Sachsenmaier M, Hinz U, Schneider L, Michalski CW, Springfeld C, Strobel O, Jager D, Ulrich A, Buchler MW. Locally Advanced Pancreatic Cancer: Neoadjuvant Therapy With Folfirinox Results in Resectability in 60% of the Patients. Ann Surg. 2016 Sep;264(3):457-63. doi: 10.1097/SLA.0000000000001850. PMID 27355262

DOCUMENTS (1):
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05132504/ICF_000.pdf